CLINICAL TRIAL: NCT03369912
Title: A Multicenter, Randomized, Patient, Investigator and Sponsor Blinded, Placebo-controlled Phase II Study to Evaluate the Efficacy and Safety of CSJ148 in Pregnant Women With Primary HCMV Infection
Brief Title: A Study to Evaluate CSJ148 in Pregnant Women With Primary HCMV Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to withdraw before study started
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCSJ148X2202; 2017-002047-15 (EudraCT Number)
Record Dates: First submitted 2017-11-28; First posted 2017-12-12 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: HCMV Infection
Keywords: Safety, efficacy; pregnant women; CSJ148; HCMV infection; congenital HCMV
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: This is a randomized, patient, investigator and sponsor blinded, placebo-controlled study in pregnant women with primary HCMV infection. This study is a non-confirmatory trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a patient, investigator and sponsor-blinded study. Patients, investigators and sponsor will remain blinded to study treatment throughout the study.
  With the exception of any unblinded site staff identified below, all site staff (including study investigator and study nurse) will be blinded to study treatment throughout the study.
  Drug product will be supplied in patient specific kits, so an unblinded pharmacist who is independent of the study team will be required in order to maintain the blind. Appropriate measures must be taken by the unblinded pharmacist to ensure that the treatment assignments are concealed from the rest of the site staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): CSJ148
  Interventions: Biological: CSJ148
- Placebo (Placebo Comparator): 5% dextrose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CSJ148 — Active
  Arms: Active
Other: Placebo — No Drug
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the feasibility of using CSJ148 to prevent congenital human cytomegalovirus (HCMV) in pregnant women with primary HCMV infection.

DETAILED DESCRIPTION:
This is a randomized, patient, investigator and sponsor blinded, placebo-controlled study in pregnant women with primary HCMV infection. The study has three periods: (I) screening (II) double-blinded placebo-controlled treatment and (III) post-delivery follow-up of women and neonates/infants. Pregnant women with confirmed primary HCMV infection will participate in periods I and II. Mothers and neonates/infants born to mothers enrolled in the study will participate in period III.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Pregnant women ≥ 18 years of age with primary HCMV infection occurring between 6 and 24 weeks of gestation
3. Ability to receive study drug within 6 weeks of the presumed onset of primary maternal infection.
4. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Confirmed or suspected fetal HCMV infection, defined as positive HCMV DNA in amniotic fluid or fetal ultrasound abnormalities suggestive of fetal HCMV disease.
2. Prior treatment with any of the following within 30 days prior to enrollment: ganciclovir, valganciclovir, foscarnet, cidofovir, acyclovir (>25 mg/kg/day IV), valacyclovir (>3 gm/day oral), famciclovir (>1500 mg/day oral), HCMV immune globulin, immune globulin (>500 mg/kg), or any other medication with anti-HCMV activity.
3. Any surgical or medical condition (other than pregnancy) which might increase the risk for thrombotic events if the patient is given immune-globulins. These conditions include cryoglobulinemia, monoclonal gammopathies, and hypertriglyceridemia (fasting level >1000 mg/dL). The investigator should make this determination based on the patient's medical history and laboratory data.
4. History of chronic hepatitis B, hepatitis C and human immunodeficiency virus (HIV) infection. Cured hepatitis C in not considered exclusionary.
5. Patient request for medical interruption or termination of pregnancy before inclusion.
6. Any surgical or medical condition which may jeopardize the patient or fetus in case of participation in the study. The investigator should make this determination in consideration of the patient's obstetrical history.
7. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer; or longer if required by local regulations.
8. History of hypersensitivity to any of the study treatments or excipients or to drugs of similar chemical classes.
9. Body weight > 100 kilograms.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant Women
Enrollment: 0 (Actual)
Dates: Start 2018-10-23 (Estimated); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Event rate of fetuses or neonates with congenital human cytomegalovirus (HCMV) infection | Day 218
  To assess the efficacy of CSJ148 on reducing intrauterine HCMV transmission compared to placebo

SECONDARY OUTCOMES:
Change from Baseline in the Reduction in symptomatic congenital human cytomegalovirus (HCMV) disease (compared to placebo) | Day 218
  Change in symptomatic HCMV disease, assessed by event rates in patients vs controls
Change from baseline in congenital human cytomegalovirus (HCMV) urine viral load in neonates at birth | Baseline, Day 218
  Change in HCMV urine viral load in neonates at birth
Pharmacokinetic concentration data of CSJ148 | Days 1,29,57,85,218,141,169, 197, 218
  Concentration of CSJ148 (LJP538 and LJP539) in serum
CSJ148 concentration in cord blood | Day 218
  Concentration of CSJ148 (LJP538 and LJP539) in serum separated from cord blood
Immunogenicity of CSJ148 in pregnant women | Days 1,29,57,85,218,141,169, 197, 218
  Detection of anti-LJP538 and anti-LJP539 antibodies in serum at selected timepoints
Immunogenicity of CSJ148 in cord blood | Day 218
  Detection of anti-LJP538 and anti-LJP539 antibodies in serum from cord blood
CSJ148 concentration in amniotic fluid | Day 218
  Concentration of CSJ148 (LJP538 and LJP539) in amniotic fluid

IPD SHARING:
Plan to Share IPD: No